CLINICAL TRIAL: NCT04114942
Title: PEERS© for Careers: An Evidence-based Social Skills Treatment for Post-secondary Employment
Brief Title: PEERS© for Careers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Amanda Gulsrud, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 11934
Record Dates: First submitted 2019-09-25; First posted 2019-10-03 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: young adult; college; transitions; career development; social skills
MeSH Terms: conditions — Autism Spectrum Disorder; Social Skills

STUDY DESIGN:
Intervention Model Description: A sequential multiple assignment randomized trial (SMART) will be conducted, with data collected at 4 major time points (baseline, post P1 (20 weeks), post P2 (10 weeks), 10-week follow up). After baseline assessments, participants will be randomized to receive the 20-week didactic training either with the assistance of a career coach or without (Phase 1). In Phase 2, individuals randomized to the coach condition will continue in the internship phase with a coach. Individuals randomized to the no-coach condition will be re-randomized to either receive assistance from a career coach during their 10-week internship or complete the internship alone. A follow-up, 10-weeks post internship, will be conducted to measure maintenance of treatment gains.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Constant Coach (Experimental): Randomized to have coach during didactic training and internship.
  Interventions: Behavioral: Constant Coach
- Internship Only Coach (Experimental): Randomized to have coach during internship only.
  Interventions: Behavioral: Internship Only Coach
- Never Coach (Experimental): Randomized to never have coach.
  Interventions: Behavioral: Never Coach

INTERVENTIONS:
Behavioral: Never Coach — 20 weeks of didactic training and 10 weeks of internship, but no coaching.
  Arms: Never Coach
Behavioral: Internship Only Coach — 20 weeks of didactic training with no coaching and 10 weeks of internship with coaching.
  Arms: Internship Only Coach
Behavioral: Constant Coach — 20 weeks of didactic training and 10 weeks of internship, with coaching throughout.
  Arms: Constant Coach

SUMMARY:
The current study proposes to investigate the effectiveness of PEERS© adapted to target postsecondary students with ASD as they prepare for careers (PEERS© for Careers). Building upon the PEERS© evidence base, PEERS© for Careers will target the development of social competence and related skills as they pertain to the work setting in a 20-week didactic course and subsequent 10-week internship. In the first phase of the study, participants will be randomized to be paired with a career coach to support practicing and generalizing the skills learned within the didactics portion of the program or to receive the didactic training without a career coach. In the second phase of the study, participants who were randomized to receive the didactic training with a coach will continue to receive coaching during the following 10-week internship phase. Those who completed the didactic training without a coach will be re-randomized to either a career coach or no coach condition and will complete a 10-week internship as well.

DETAILED DESCRIPTION:
Young adults with autism spectrum disorder (ASD) often experience poor postsecondary employment outcomes; significantly worse than would be expected based upon their cognitive abilities. Social skills deficits are a major contributor to the challenges young adults with ASD experience obtaining and maintaining employment. Across studies, research indicates rates of unemployment from 40 to 75% for the ASD population, compared to 18.5% for the general population of young adults in the same year. Data from a nationally representative survey of young adults indicated that only 53.4% of individuals with ASD had ever worked for pay since high school, and only 33.6% were currently employed. This reflects a rate of unemployment that is four times higher than individuals with intellectual disability, and six to 12 times higher than individuals with prior special education services under categories other than "Autism," even after adjusting for covariates such as adaptive skills and conversational ability.

Despite this substantial gap in employment attainment for individuals with ASD, there are limited services available to support the transition from post-secondary education to the workforce. Existing services often focus on vocational training and supports, rather than underlying social skill deficits, and are typically designed for individuals with comorbid intellectual disabilities. Recently, a randomized control trial was conducted using the Project SEARCH intervention, which was modified for high school seniors with ASD. Results were promising, including higher rates of job attainment and higher wages after the intervention.

It is clear that additional intervention development and rigorous research is needed to address the ASD employment gap, particularly for individuals who have completed high school and have age-typical intellectual abilities. The Program for the Education and Enrichment of Relational Skills (PEERS©) is one of the only evidence-based social skills interventions for adolescents and adults with ASD. PEERS© has been disseminated world-wide with consistent positive outcomes that are maintained over time, including improvements in social responsiveness, cooperation, and self-control, as well as increased frequency of peer get-togethers and a reduction in ASD-related mannerisms and preoccupations.

While social skills interventions have helped young adults with ASD improve friendship skills, there is a paucity of comprehensive evidence-based treatments focused on the social skills young adults need to obtain and maintain employment. The success of the PEERS© program in improving friendship-related social skills, coupled with the significant employment challenges experienced by this population, was the impetus for the development of the comprehensive employment transition program PEERS© for Careers.

The current study proposes to investigate the effectiveness of PEERS© adapted to target postsecondary students with ASD as they prepare for careers (PEERS© for Careers). Building upon the PEERS© evidence base, PEERS© for Careers will target the development of social competence and related skills as they pertain to the work setting in a 20-week didactic course and subsequent 10-week internship. In the first phase of the study, participants will be randomized to be paired with a career coach to support practicing and generalizing the skills learned within the didactics portion of the program or to receive the didactic training without a career coach. In the second phase of the study, participants who were randomized to receive the didactic training with a coach will continue to receive coaching during the following 10-week internship phase. Those who completed the didactic training without a coach will be re-randomized to either a career coach or no coach condition and will complete a 10-week internship as well.

ELIGIBILITY:
Inclusion Criteria - Participants will be eligible if they meet the following criteria:

* graduated from high school (GED or diploma)
* between the ages of 18-35
* currently or have history of enrollment in post-secondary education (e.g. junior college, community college, 4-year university)
* have a pre-existing ASD diagnosis without severe co-morbid mental health disorders that may actively impair their ability to participate in the PEERS© for Careers program (e.g., psychosis)
* have intellectual functioning at or above the average range (>85).

Exclusion Criteria - Participants will NOT be eligible if they:

* have not graduated from high school (GED or diploma)
* are not between the ages of 18-35
* are not currently of have a history of enrollment in post-secondary education (e.g. junior college, community college, 4-year university)
* do not have a pre-existing ASD diagnosis, or they have a severe co-morbid mental health disorders that may actively impair their ability to participate in the PEERS© for Careers program (e.g., psychosis)
* have intellectual functioning below the average range (<85).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Change in Employment-related Social Skills Knowledge as Assessed by Test of Employment Social Skills (TESS) | baseline (entry), after 20-week didactic (20 weeks after entry), after 10-week internship (30 weeks after entry), at 10-week follow-up (40 weeks after entry)
  The Test of Employment Social Skills (TESS) is a novel, 36-item criterion-referenced measure created to assess young adults' knowledge of the specific social and employment-related skills taught during the intervention. Changes from baseline in TESS scores after 20-week didactic, 10-week internship, and 10-week follow-up will be compared across different interventions.
Change in Employment-related Social Skills Knowledge as Assessed by Adapted Contextual Assessment of Social Skills (CASS) | baseline (entry), after 20-week didactic (20 weeks after entry), after 10-week internship (30 weeks after entry), at 10-week follow-up (40 weeks after entry)
  The Contextual Assessment of Social Skills (CASS) is a role-play assessment of conversational skills for verbally-fluent adolescents and young adults with ASD which is systematically behaviorally coded. The CASS will be adapted for a work-setting scenario. Change from baseline in CASS scores after 20-week didactic, 10-week internship, and 10-week follow-up will be compared across different interventions.
Change in Social Skills Knowledge as Assessed by Social Responsiveness Scale (SRS-2) | baseline (entry), after 20-week didactic (20 weeks after entry), after 10-week internship (30 weeks after entry), at 10-week follow-up (40 weeks after entry)
  The Social Responsiveness Scale (SRS-2) is a standardized, validated measure of severity of ASD symptoms as they occur in natural settings. Changes from baseline in SRS-2 scores after 20-week didactic, 10-week internship, and 10-week follow-up will be compared across different interventions.

SECONDARY OUTCOMES:
Autism Severity as Assessed by Wechsler Abbreviated Scale of Intelligence (WASI-II) | baseline (entry)
  The Wechsler Abbreviated Scale of Intelligence (WASI-II) is a standardized, abbreviated measure of cognitive ability. Scores on the WASI-II at baseline will be analyzed to test whether autism severity at baseline moderates the effect of the intervention as assessed by changes in TESS, CASS, and SRS-2 scores.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda C Gulsrud, PhD, Principal Investigator — University of California, Los Angeles; Elizabeth A Laugeson, PsyD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA CAN Clinic, Los Angeles, California
  - UCLA PEERS Clinic, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laugeson EA, Gantman A, Kapp SK, Orenski K, Ellingsen R. A Randomized Controlled Trial to Improve Social Skills in Young Adults with Autism Spectrum Disorder: The UCLA PEERS((R)) Program. J Autism Dev Disord. 2015 Dec;45(12):3978-89. doi: 10.1007/s10803-015-2504-8. PMID 26109247
- [Background] Ohl A, Grice Sheff M, Small S, Nguyen J, Paskor K, Zanjirian A. Predictors of employment status among adults with Autism Spectrum Disorder. Work. 2017;56(2):345-355. doi: 10.3233/WOR-172492. PMID 28211841
- [Background] Roux AM, Shattuck PT, Cooper BP, Anderson KA, Wagner M, Narendorf SC. Postsecondary employment experiences among young adults with an autism spectrum disorder. J Am Acad Child Adolesc Psychiatry. 2013 Sep;52(9):931-9. doi: 10.1016/j.jaac.2013.05.019. Epub 2013 Jul 31. PMID 23972695
- [Background] Taylor JL, Seltzer MM. Employment and post-secondary educational activities for young adults with autism spectrum disorders during the transition to adulthood. J Autism Dev Disord. 2011 May;41(5):566-74. doi: 10.1007/s10803-010-1070-3. PMID 20640591